CLINICAL TRIAL: NCT00586625
Title: Safety Study for Bepotastine Besilate Ophthalmic Solution in Normal Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-SAF-0405071-P
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2009-11-11 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — bepotastine besilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bepreve (Experimental): bepotastine besilate ophthalmic solution 1.5%
  Interventions: Drug: Bepreve
- Placebo (Placebo Comparator): vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bepreve — One drop, both eyes, twice a day
  Arms: Bepreve
Drug: Placebo — One drop, both eyes, twice a day
  Arms: Placebo

SUMMARY:
Safety study for bepotastine besilate ophthalmic solution in normal volunteers

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 3 years of age, and have ocular health within normal limits

Exclusion Criteria:

* No active ocular disease

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5%; Placebo (Vehicle): One drop, both eyes, twice a day for six weeks
Period: Overall Study
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo (Vehicle)
Started | 575 | 286
Completed | 532 | 269
Not Completed | 43 | 17
Not completed — Adverse Event | 6 | 6
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 32 | 10
Not completed — Subject non-compliance | 0 | 1
Not completed — Subject unable to return for visit | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo (Vehicle) | Total
Number analyzed (Participants) | 575 | 286 | 861
Age, Customized [Number; unit: participants]
  3-9 years | 47 | 25 | 72
  10-17 years | 40 | 15 | 55
  >=18 years | 488 | 246 | 734
Age Continuous [Mean (Standard Deviation); unit: years] | 34.5 (16.5) | 34.2 (16.3) | 34.4 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367 | 178 | 545
  Male | 208 | 108 | 316

OUTCOME MEASURES:

1. Primary Outcome: Ocular Comfort
Description: A 4-step grading scale with half unit (1-step) increments allowed:
  0=Comfortable;discomfort absent; 1.0=Generally comfortable; mild discomfort; 2.0=Some discomfort but tolerable; moderate comfort; 3.0=Severely uncomfortable or intolerable
Time Frame: Day 8 & Day 22
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo (Vehicle)
Number analyzed (Participants) | 575 | 286
Scores on a scale
  Day 8: Upon instillation | 0.13 (0.35) | 0.07 (0.26)
  Day 8: 5 minutes after instillation | 0.06 (0.25) | 0.02 (0.13)
  Day 22: Upon instillation | 0.1 (0.33) | 0.06 (0.23)
  Day 22: 5 minutes after instillation | 0.05 (0.22) | 0.04 (0.17)

ADVERSE EVENTS:
Arm/Group | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% | Placebo (Vehicle)
Serious Adverse Events (participants affected / at risk) | 0/575 | 0/286
Other Adverse Events (participants affected / at risk) | 146/575 | 7/286
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bepreve (Bepotastine Besilate Ophthalmic Solution) 1.5% (N=575) | Placebo (Vehicle) (N=286)
Mild Taste (Nervous system disorders) | 146 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement is between contract research organization and third parties on behalf of ISTA Pharmaceuticals, Inc.